CLINICAL TRIAL: NCT00787020
Title: Ventriculostomies in SAH: ICP Open or Not?
Acronym: VISION
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00005900
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Results first posted 2010-12-17 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2011-03

CONDITIONS: Subarachnoid Hemorrhage
Keywords: Cerebrospinal Fluid; Ventriculostomy; Subarachnoid hemorrhage; vasospasm; Human Subjects
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ventriculostomy Open: Subjects are treated with near continuous cerebrospinal fluid (CSF) diversion by positioning the stopcock in the open position and the intracranial pressure (ICP) is monitored once each hour: CSF drains into an external ventricular drainage bag.
- Ventriculostomy Monitored: Subjects are treated with intermittent cerebrospinal fluid (CSF) diversion. Intracranial pressure (ICP) is monitored and CSF is drained only when the ICP exceeds a threshold dictated by the attending physician.

SUMMARY:
The purpose of this study is explore how cerebrospinal fluid (CSF) drainage impacts outcomes for patients diagnosed with subarachnoid hemorrhage (SAH). This is a non-randomized observational study of two physician-prescribed approaches to managing intracranial pressure monitoring and CSF drainage for SAH patients. The study will enroll only those patients who have intracranial pressure (ICP) monitoring in situ. Because this is an observational study, there are no physical risks to the patient, the only risk is loss of confidentiality.

DETAILED DESCRIPTION:
There are no interventions specific to this observational study. The nurses and physicians who care for subjects in the study are already competent in the care and management of patients with subarachnoid hemorrhage (SAH) and intracranial pressure (ICP) monitoring as a requirement of their current employment at Duke University. Patients with confirmed diagnosis of subarachnoid hemorrhage requiring ICP and CSF management will be admitted to the 16 bed Neurocritical Care Unit (NCCU) at Duke Hospital. After admission procedures and a baseline neurologic assessment are complete, the charge nurse or NCCU fellow will notify an investigator of subjects meeting inclusion criteria. The investigator or research coordinator for this project will complete a review preparatory to research (RPR) to ensure no exclusion criteria are present and once subject appropriateness has been confirmed patients and their families will be introduced to the investigator for the purpose of obtaining informed consent. The subject's legally authorized representative (LAR) will be informed of the study's purpose, risks and benefits, and the rights of research subjects.

Data will be collected that reflects the duration of the patient's hospitalization at Duke University through chart abstraction. The study period will be defined as admission to discharge. The attending physician has, and will continue to, determine the appropriateness of the duration of ICP monitoring, NCCU discharge criteria and hospital discharge criteria. Chart abstraction will be completed daily to obtain the ICP values and CSF volumes during that period of time for which the patient has a ventriculostomy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of subarachnoid hemorrhage
* Age 18 years or older
* Ventriculostomy in situ

Exclusion Criteria:

* Prisoners
* Glasgow coma score = 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subarachnoid hemorrhage
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2008-11; Primary Completion 2009-08 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: DaiWai M Olson, PhD RN, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

REFERENCES:
- [Result] Kim GS, Amato A, James ML, Britz GW, Zomorodi A, Graffagnino C, Zomorodi M, Olson DM. Continuous and intermittent CSF diversion after subarachnoid hemorrhage: a pilot study. Neurocrit Care. 2011 Feb;14(1):68-72. doi: 10.1007/s12028-010-9401-y. PMID 20596794

RESULTS

PARTICIPANT FLOW:
Groups:
- Ventriculostomy Open: Subjects are treated with near continuous cerebrospinal fluid (CSF) diversion by position the stopcock in the open position and the intracranial pressure (ICP) is monitored each hour: CSF drains into an external ventricular drainage bag.
Period: Overall Study
Arm/Group | Ventriculostomy Open | Ventriculostomy Monitored
Started | 24 | 13
Completed | 24 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ventriculostomy Open | Ventriculostomy Monitored | Total
Number analyzed (Participants) | 24 | 13 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 10 | 30
  >=65 years | 4 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.92 (13.35) | 53.13 (11.13) | 54.11 (11.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 9 | 25
  Male | 8 | 4 | 12
Region of Enrollment [Number; unit: participants]
  United States | 24 | 13 | 37

OUTCOME MEASURES:

1. Primary Outcome: Cerebral Artery Vasospasm
Description: Cerebral artery vasospasm is defined as transcranial doppler mean velocity greater than 120 or angiographic vasospasm determined by cerebral angiogram.
Time Frame: 14 days
Measure: Number; unit: Participants
Arm/Group | Ventriculostomy Open | Ventriculostomy Monitored
Number analyzed (Participants) | 24 | 13
Participants | 16 | 7

2. Secondary Outcome: External Ventricular Drain (EVD) Complications
Description: External ventricular drain complications are defined as ventriculitis, shunt dependency, ventricular catheter obstruction requiring manipulation, or removal by the patient.
Time Frame: 14 Days
Measure: Number; unit: Participants
Arm/Group | Ventriculostomy Open | Ventriculostomy Monitored
Number analyzed (Participants) | 24 | 13
Participants | 14 | 4

3. Secondary Outcome: Cerebrospinal Fluid (CSF) Output Per Day
Time Frame: 14 Days
Measure: Mean (95% Confidence Interval); unit: Milliliter
Arm/Group | Ventriculostomy Open | Ventriculostomy Monitored
Number analyzed (Participants) | 24 | 13
Milliliter | 134 [116.9 to 151.1] | 135 [112.2 to 157.8]

ADVERSE EVENTS:
Arm/Group | Ventriculostomy Open | Ventriculostomy Monitored
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/13
Other Adverse Events (participants affected / at risk) | 0/24 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No